CLINICAL TRIAL: NCT05053633
Title: Relationship Between Analgesia Nociception Index, Anxiety, and Pain in Conscious Hernia Patients Undergoing Combined Spinal Epidural Anesthesia
Brief Title: Relationship Between ANI, Anxiety, and Pain in Conscious Hernia Patients Undergoing CSEA
Status: Completed | Type: Observational
Sponsor: Beijing Chao Yang Hospital (Other)
Responsible Party: Principal Investigator, Changwei Wei, Deputy chief physician, Beijing Chao Yang Hospital
Other Study IDs: 00375931
Record Dates: First submitted 2021-09-15; First posted 2021-09-22 (Actual); Last update posted 2024-08-13 (Actual); Status verified 2024-08

CONDITIONS: Combined Spinal-epidural Anesthesia

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Combined spinal epidural anesthesia: The assessments are conducted in conscious patients under the procedure of Combined spinal epidural anesthesia.
  Interventions: Procedure: Combined spinal epidural anesthesia

INTERVENTIONS:
Procedure: Combined spinal epidural anesthesia — The Anxiety (Visual Analogue Scale for Anxiety), pain (Visual Analogue Scale), and the Analgesia Nociception Index (ANI) assessments are conducted at four specific time points: lateral position, local anesthesia, epidural needle puncture and 2 minutes after puncture.

SUMMARY:
Analgesia Nociception Index can be used to detect noxious stimulation during general anesthesia.The aim of this study is to observe ANI under combined spinal epidural anesthesia procedures in conscious hernia patients.

DETAILED DESCRIPTION:
Analgesia Nociception Index which is derived by heart rate variability, can be used to detect noxious stimulation during general anesthesia. However, the impact of anxiety on ANI evaluation and the correlation between ANI, pain, and anxiety in awake patients remains unclear. This study aimed to investigate the correlation between ANI, pain, and anxiety in conscious hernia patients undergoing combined spinal epidural anesthesia procedures.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18- 80 years
* ASA physical status I or II
* Scheduled for inguinal hernia, umbilical hernia or incisional repair under CSEA
* Written informed consent

Exclusion Criteria:

* Use of CNS-active medication or abuse of alcohol
* History of cardiac arrhythmia
* Contraindications of combined spinal epidural anesthesia
* Previous exposure to CSEA or surgery

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants with ASA status I or II, aged between 18 and 80 years old, scheduled for inguinal hernia, umbilical hernia or incisional repair under CSEA were included in the study. Participants with chronic pain, cardiovascular dysfunction, arrhythmia, dysautonomia, pacemaker usage, medication affecting the autonomic nervous system, contraindications to CSEA, or previous exposure to CSEA or surgery were excluded.
Sampling Method: Probability Sample
Enrollment: 24 (Actual)
Dates: Start 2021-09-25 (Actual); Primary Completion 2023-02-25 (Actual); Study Completion 2023-05-31 (Actual)

PRIMARY OUTCOMES:
The correlation between ANI and pain (measured with Visual Analog Scale,VAS), ANI and anxiety (measured with Visual Analog Scale-Anxiety,VAS-A) changes in conscious patients during anesthesia procedures | The changes of ANI, VAS, and VAS-A, from baseline at different Time-points to 2min after anesthesia procedures, (Timepoints: T1=after lateral position, T2=local anesthesia, T3=epidural needle puncture, and T4=2 minutes after puncture)
  ANI is derived from hear rate variability, ranging from 0-100, bigger number means better analgesic level. Patients undergoing CSEA may experience mid-level anxiety while remaining conscious. The anxiety (VAS-A), pain (VAS), and ANI assessments were conducted at four specific time points.

SECONDARY OUTCOMES:
The correlation between pain (measured with Visual Analog Scale,VAS) and anxiety (measured with Visual Analog Scale-Anxiety,VAS-A) changes in conscious patients during anesthesia procedures | The changes of VAS, and VAS-A, from baseline at different Time-points to 2min after anesthesia procedures, (Timepoints: T2=local anesthesia, T3=epidural needle puncture, and T4=2 minutes after puncture)
  The anxiety (VAS-A) and pain (VAS) were conducted at three specific time points, since there is no stimulus at lateral position (Timepoints: T2=local anesthesia, T3=epidural needle puncture, and T4=2 minutes after puncture).

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Chao Yang Hospital, Beijing, Beijing Municipality, China